CLINICAL TRIAL: NCT07152041
Title: A Phase 3, Multicenter Trial for Pediatric Philadelphia Chromosome-positive B-Acute Lymphoblastic Leukemia -2025 Project
Brief Title: Newly-diagnosed Pediatric Ph-positive B-ALL Protocol
Acronym: CAMS-Ph+ B-ALL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025041
Record Dates: First submitted 2025-03-28; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia (ALL) Philadelphia Chromosome-positive (Ph+); Childhood Leukemia, Acute Lymphoblastic
Keywords: olverembatinib; Blinatumomab; venetoclax
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — olverembatinib; Vincristine; Prednisone; blinatumomab; Methotrexate; Cytarabine; Daunorubicin; venetoclax; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OVB+Blina+VEN+Chemo-light regimen (Experimental): All Ph+-ALL patients will uniformly use the 3rd generation of TKI olverembatinib (OVB) instead of dasatinib throughout the regimen. Cyclophosphamide and asparaginase are totally omitted from the entire treatment to mitigate toxicities.
  OVB is combined with Vincristine and Prednisone (VP) during the first 2 weeks and with blinatumomab during the last 4 weeks of remission induction in this protocol.
  Patients will receive blinatumomab for 28 days as induction instead of CAT to improve induction response and avoid toxicity.
  All patients will receive two cycles of HDMTX+Blina-14 and 4 times of triple intrathecal therapy (TIT) throughout the consolidation 1 phase. The dosage of AraC will be reduced to 1 g/m2 in the consolidation 2 phase.
  Throughout the early Maintenance Therapy, dexamethasone and vincristine combination will be added with either venetoclax or daunorubicin alternatively for five cycles, given after MTX and 6-MP.
  Interventions: Drug: olverembatinib

INTERVENTIONS:
Drug: olverembatinib — All Ph+-ALL patients will uniformly use the 3rd generation of TKI olverembatinib (OVB) instead of dasatinib throughout the regimen.
  OVB is combined with Vincristine and Prednisone (VP) during the first 2 weeks and with blinatumomab during the last 4 weeks of remission induction in this protocol.
  Patients will receive blinatumomab for 28 days as induction instead of CAT to improve induction response and avoid toxicity.
  All patients will receive two cycles of HDMTX+Blina-14 and 4 times of triple intrathecal therapy (TIT) throughout the consolidation 1 phase.
  To decrease the toxicities of high-dose AraC, the dosage will be reduced to 1 g/m2 in the consolidation 2 phase in contrast to 2 g/m2 in 2020 protocol.
  Throughout the early Maintenance Therapy, dexamethasone and vincristine combination will be added with either venetoclax or daunorubicin alternatively for five cycles, given after MTX and 6-MP.
  Other Names: vincristine; prednisone; blinatumomab; Methotrexate; Cytarabine; Daunorubicin; venetoclax; Dexamethasone; 6-MP

SUMMARY:
This prospective clinical trial evaluates the effectiveness and safety of "chemotherapy-light" regimen incorporating the third-generation TKI olverembatinib, the bi-specific CD3/CD19 T cell engager blinatumomab, and the BCL-2 selective inhibitor venetoclax for newly diagnosed pediatric/adolescent patients with Ph+ ALL. The CCCG-Ph+ B-ALL-2025 protocol will be modified as following compared to the CCCG-ALL-2020 protocol

DETAILED DESCRIPTION:
1. All Ph+-ALL patients will uniformly use the 3rd generation of TKI olverembatinib (OVB) instead of dasatinib throughout the regimen.
2. OVB is combined with Vincristine and Prednisone (VP) during the first 2 weeks and with blinatumomab during the last 4 weeks of remission induction in this protocol.
3. Patients will receive blinatumomab for 28 days as induction instead of CAT to improve induction response and avoid toxicity.
4. All patients will receive two cycles of HDMTX+Blina-14 and 4 times of triple intrathecal therapy (TIT) throughout the consolidation 1 phase.
5. To decrease the toxicities of high-dose AraC, the dosage will be reduced to 1 g/m2 in the consolidation 2 phase in contrast to 2 g/m2 in 2020 protocol.
6. Throughout the early Maintenance Therapy, dexamethasone and vincristine combination will be added with either venetoclax or daunorubicin alternatively for five cycles, given after MTX and 6-MP.
7. Cyclophosphamide and asparaginase are totally omitted from the entire treatment to mitigate toxicities.
8. Olverembatinib concentrations are recommended to be examined (cerebrospinal fluid and peripheral blood in parallel) before OVB given, after full dosing of OVB, and/or Blina+OVB, best to match lumbar puncture assessments timepoints.
9. IgH rearrangement by NGS MRD will be added as an evaluation indicator, with testing frequency matching bone marrow aspiration assessments.
10. Pharmarcotyping studies are recommended at baseline if condition permits.
11. For patients who cannot use full-dose blinatumomab, we will adopt the CCCG-Ph+ALL2020 protocol. complications.

ELIGIBILITY:
Inclusion Criteria:

Must meet all items below:

1. Age older than 1 month to younger 18 years.
2. Newly diagnosed Philadelphia chromosome-positive or BCR::ABL1-positive B-ALL.
3. Written informed consent of the parents or other legally authorized guardian of the patient according to local law and regulations.

Exclusion Criteria:

Should be excluded if had any item below:

1. ALL evolved from CML.
2. Known underlying congenital immunodeficiency or metabolic disease.
3. Congenital heart disease with cardiac insufficiency.
4. Gastrointestinal dysfunction or gastrointestinal diseases that may significantly alter the absorption of study drug.
5. Severe malnutrition, uncontrolled active infections, or serious cardiovascular diseases.
6. Subjects with significant CNS disorder (e.g., uncontrolled seizure disorder, autoimmune disease involving CNS).
7. Treated with glucocorticoids for ≥14 days, or targeted inhibitor for > 7 days within one month before enrollment, or any chemotherapy or any systemic anticancer therapy (including but not limited to any TKI) or radiotherapy within 3 months before enrollment (except for emergency radiotherapy to relieve airway compression).
8. Any significant comorbidities or psychiatric disorders that may impact patient safety, compliance, informed consent, study participation, follow-up, or the interpretation of study results. In such cases, all participating sites must report directly to the PI to determine whether the patient meets exclusion criteria.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Day 48 end-of-induction measurable residual diseases (MRD48) after induction remission with olverembatinib and blinatumomab, compared to MRD46 of those treated with dasatinib plus chemotherapy induction (CCCG-ALL-2015 /2020) or from historical cohorts . | Up to approximately 4.5 years.
  Primary analysis will be performed by one-sided (Monte-Carlo-) exact chi-square test because the objective calls for testing if the proportion of patients in the <0.01% Day 48 MRD group is higher than the historical control. The historical control of Day 46 MRD of dasatinib combination with intensive chemotherapy is 80%. It is estimated that VPO+Blinatumomab can increase the negative rate of Day 48 MRD by 10%. a total sample size of 135 provides sufficient power for the planned analyses outlined above if the true D48 MRD negativity probability is 0.90 or higher based on a one-sided alpha of 0.05.

SECONDARY OUTCOMES:
Day 19 measurable residual diseases (MRD19) during induction remission with olverembatinib plus VP (VOP), compared to MRD19 of those treated with dasatinib plus 4-drug chemotherapy induction (CCCG-ALL-2015 /2020) or from historical cohorts | Approximately 4.5 years.
  For this objective a one-sided comparison of probabilities and historical control rate of 40% will be made. Let p2 be the probability of achieving negative D19 MRD on the current study, then the one-sided alternative hypothesis H0: p2=40% vs. H1: p2>40% will be tested. This analysis will be performed by one-sample one-sided exact binomial test, based on a one-sided alpha of 0.025. The historical control is based on the MRD of patients treated on CCCG-ALL-2015.
Event-free survival (EFS) of patients treated with this therapy, in comparison to historical regimens. | Approximately 7 years.
  The EFS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 2, 3 years since diagnosis). Standard error will be estimated using the default procedure in R. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of EFS will be performed using two-sided log-rank test. Multivariable regression modeling including trial (CAMS-Ph+B-ALLRegimen 2025 vs. CCCG-Ph-ALL 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
Overall survival (OS) of patients treated with this therapy, in comparison to historical regimens | Approximately 7 years.
  The OS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 2, 3 years since diagnosis). Comparison of OS functions will be conducted using the two-sided log-rank test. Standard error will be estimated using the default procedure in R. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of OS will be performed using two-sided log-rank test. Multivariable regression modeling including trial (CAMS-Ph+B-ALL-2025 vs. CCCGALL-2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
Cumulative incidence of relapse (CIR) of this therapy, in comparison to historical regimens. | Approximately 7 years.
  CIR functions of relapse will be estimated by the Kalbafleisch-Prentice method. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of CIR will be performed by Gray's test. Multivariable regression modeling including trial (CAMS-Ph+B-ALLALL-2025 vs. CCCGALL-2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Fine-Gray models.

OTHER OUTCOMES:
To correlate measurable residual diseases (MRD) during remission induction and after consolidation by Ig-NGS, qPCR of BCR::ABL1 and FCM-MRD with cumulative incidence of event-free survival (EFS) | Approximately 7 years
  Proportions of patients with positive MRD by NGS, qPCR and FCM on Days 19 and 48 will be estimated by the sample proportion along with the 95% confidence interval. The EFS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 2 3 years since diagnosis). Comparisons of OS and EFS will be done by log-trank test, and comparison of CIR will be done by Gray's test. Multivariable regression modeling including trial (CAMS-Ph+B-ALL-2025 vs. CCCGALL-2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
To correlate measurable residual diseases (MRD) during remission induction and after consolidation by Ig-NGS, qPCR of BCR::ABL1 and FCM-MRD with cumulative incidence of relapse(CIR) | Approximately 7 years
  Proportions of patients with positive MRD by NGS, qPCR and FCM on Days 19 and 48 will be estimated by the sample proportion along with the 95% confidence interval. The CIR curve will be estimated by Kalbafleisch-Prentice method, along with 95% confidence intervals at specified timepoints (e.g., 2 3 years since diagnosis). Comparisons of CIR will be done by Gray's test. Multivariable regression modeling including trial (CAMS-Ph+B-ALL-2025 vs. CCCGALL2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Fine-Gray models(CIR).
To correlate measurable residual diseases (MRD) during remission induction and after consolidation by Ig-NGS, qPCR of BCR::ABL1 and FCM-MRD with overall survival (OS) | Approximately 7 years
  Proportions of patients with positive MRD by NGS, qPCR and FCM on Days 19 and 48 will be estimated by the sample proportion along with the 95% confidence interval. The OS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 2 3 years since diagnosis). Comparisons of OS will be done by log-rank test. Multivariable regression modeling including trial (CAMS-Ph+B-ALL-2025 vs. CCCGALL-2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
Incidence of Grade 3 or higher Treatment-Emergent Adverse Events (TEAE) associated with olverembatinib, venetoclax and blinatumomab, and compared with the historical controls treated with dasatinib plus intensive chemotherapy. | Up to 30 days after last dose of study treatment
  Proportions of grade-3 or higher TEAEs in each treatment phase will be estimated by the sample proportions along with exact 95% confidence intervals. Cumulative incidences of various grade-3 or higher AEs throughout therapy will be estimated by the Kalbafleisch-Prentice method; death, relapse and other events rendering off therapy before completion are regarded as competing risks.
To explore the relationship between cellular immunity dynamics during olverembatinib treatment and the efficacy of blinatumomab-contained therapy. | Approximately 7 years
  Descriptive statistics including correlation coefficients (Pearson's or Spearman's) and regression modeling including possibly longitudinal data models will be applied as appropriate to analyze the biological associations. Associations between cellular immunity dynamics and relapse will be analysed using Gray's test or Fine-Gray regression models, as appropriate.
To explore the pharmacokinetic profiles as Maximum Plasma Concentration [Cmax] in blood paired with cerebrospinal fluid of olverembatinib given alone and in combination with blinatumomab or with prednisone plus vincristine | Up to 30 days after last dose of study treatment
  In pharmacokinetic (PK) studies of Cmax, descriptive statistics (mean, standard deviation, median, range) will be used to summarize the data. Visualizations, such as box plots and line graphs, will be used to depict the drug's concentration over time in blood and cerebrospinal fluid. Centers with the appropriate resources may conduct these analyses.
To explore the pharmacokinetic profiles as Time to Reach Maximum Plasma Concentration (Tmax) in blood paired with cerebrospinal fluid of olverembatinib given alone and in combination with blinatumomab or with prednisone plus vincristine | Up to 30 days after last dose of study treatment
  In pharmacokinetic (PK) studies as Tmax, descriptive statistics (e.g., mean, standard deviation, five-number summary) are used to summarize the data, while visualizations like box plots and line graphs are employed to depict the drug's behavior in the body. It is recommended that centers with the appropriate resources and interest consider undertaking these studies.
To explore the pharmacokinetic profiles as Area Under the Plasma Concentration-Time Curve (AUC) in blood paired with cerebrospinal fluid of olverembatinib given alone and in combination with blinatumomab or with prednisone plus vincristine | Up to 30 days after last dose of study treatment
  In pharmacokinetic (PK) studies of AUC, descriptive statistics (e.g., mean, standard deviation, five-number summary) are used to summarize the data, while visualizations like box plots and line graphs are employed to depict the drug's behavior in the body. It is recommended that centers with the appropriate resources and interest consider undertaking these studies.
To explore the pharmacokinetic profiles as Half-Life (t½) in blood paired with cerebrospinal fluid of olverembatinib given alone and in combination with blinatumomab or with prednisone plus vincristine | Up to 30 days after last dose of study treatment
  In pharmacokinetic (PK) studies of t½, descriptive statistics (e.g., mean, standard deviation, five-number summary) are used to summarize the data, while visualizations like box plots and line graphs are employed to depict the drug's behavior in the body. It is recommended that centers with the appropriate resources and interest consider undertaking these studies.
To explore the pharmacokinetic profiles as Clearance (CL) in blood paired with cerebrospinal fluid of olverembatinib given alone and in combination with blinatumomab or with prednisone plus vincristine | Up to 30 days after last dose of study treatment
  In pharmacokinetic (PK) studies of CL, descriptive statistics (e.g., mean, standard deviation, five-number summary) are used to summarize the data, while visualizations like box plots and line graphs are employed to depict the drug's behavior in the body. It is recommended that centers with the appropriate resources and interest consider undertaking these studies.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, MD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, CAMS & PUMC
Locations (23):
- China (22):
  - Anhui Medical University Second Affiliated Hospita, Hefei, Anhui
  - Chongqing Medical University Affiliated Children's Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Children's Hospital, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of the Central South University, Changsha, Hunan
  - Nanjing Children's Hospital Affiliated to Nanjing Medical University, Nanjin, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Children's Hospital, Shanghai, Shanghai Municipality
  - Shenzhen Children's Hospital, Shenzhen, Shenzhen
  - West China Second University Hospita, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, CAMS & PUMC, Tianjin, Tianjin Municipality
- Hong Kong Children's Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
1. Demographic Data: Age, sex, and other relevant baseline characteristics.
  2. Treatment Information: Data on interventions received by participants, including dosage, treatment cycles, and duration.
  3. Outcome Measures: Detailed information on primary and secondary outcome measures, such as response rates, survival rates, adverse events, and any the pre-specified endpoints.
  4. Adverse Events: Data on all reported adverse events, including severity, duration, and outcome.
  5. Laboratory Data: Results from laboratory tests, such as blood counts, biochemical markers, or molecular analysis.
  6. Medical History: Pre-existing conditions, comorbidities, and prior treatments or interventions.
  7. Vital Signs: relevant physiological data.
  8. Efficacy and Safety Data: Any data relating to the efficacy (e.g., event-free survival) and safety (e.g., adverse effects) of the treatment.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available upon publication of the primary trial results or after trial completion, whichever occurs first, starting on 2032, and will remain accessible for 5 years.
Access Criteria: Researchers, healthcare professionals who meet the criteria for access (e.g., academic researchers conducting secondary analyses or regulatory bodies reviewing safety data) will be able to request access to de-identified IPD and supporting information. Access will be facilitated through clinical trials.gov/emailing to PI, where users can submit a request and provide a research proposal. Data access will be granted after a formal review and approval process, subject to compliance with the data-sharing agreement and confidentiality terms.
URL: https://login.imedidata.com

REFERENCES:
- [Background] Manabe A, Kawasaki H, Shimada H, Kato I, Kodama Y, Sato A, Matsumoto K, Kato K, Yabe H, Kudo K, Kato M, Saito T, Saito AM, Tsurusawa M, Horibe K. Imatinib use immediately before stem cell transplantation in children with Philadelphia chromosome-positive acute lymphoblastic leukemia: Results from Japanese Pediatric Leukemia/Lymphoma Study Group (JPLSG) Study Ph(+) ALL04. Cancer Med. 2015 May;4(5):682-9. doi: 10.1002/cam4.383. Epub 2015 Jan 31. PMID 25641907
- [Background] Hum RM, Deambrosis D, Lum SH, Davies E, Bonney D, Guiver M, Turner A, Wynn RF, Hiwarkar P. Molecular monitoring of adenovirus reactivation in faeces after haematopoietic stem-cell transplantation to predict systemic infection: a retrospective cohort study. Lancet Haematol. 2018 Sep;5(9):e422-e429. doi: 10.1016/S2352-3026(18)30130-3. PMID 30172346
- [Background] Biondi A, Schrappe M, De Lorenzo P, Castor A, Lucchini G, Gandemer V, Pieters R, Stary J, Escherich G, Campbell M, Li CK, Vora A, Arico M, Rottgers S, Saha V, Valsecchi MG. Imatinib after induction for treatment of children and adolescents with Philadelphia-chromosome-positive acute lymphoblastic leukaemia (EsPhALL): a randomised, open-label, intergroup study. Lancet Oncol. 2012 Sep;13(9):936-45. doi: 10.1016/S1470-2045(12)70377-7. Epub 2012 Aug 14. PMID 22898679
- [Background] Schultz KR, Carroll A, Heerema NA, Bowman WP, Aledo A, Slayton WB, Sather H, Devidas M, Zheng HW, Davies SM, Gaynon PS, Trigg M, Rutledge R, Jorstad D, Winick N, Borowitz MJ, Hunger SP, Carroll WL, Camitta B; Children's Oncology Group. Long-term follow-up of imatinib in pediatric Philadelphia chromosome-positive acute lymphoblastic leukemia: Children's Oncology Group study AALL0031. Leukemia. 2014 Jul;28(7):1467-71. doi: 10.1038/leu.2014.30. Epub 2014 Jan 20. PMID 24441288
- [Background] Schultz KR, Bowman WP, Aledo A, Slayton WB, Sather H, Devidas M, Wang C, Davies SM, Gaynon PS, Trigg M, Rutledge R, Burden L, Jorstad D, Carroll A, Heerema NA, Winick N, Borowitz MJ, Hunger SP, Carroll WL, Camitta B. Improved early event-free survival with imatinib in Philadelphia chromosome-positive acute lymphoblastic leukemia: a children's oncology group study. J Clin Oncol. 2009 Nov 1;27(31):5175-81. doi: 10.1200/JCO.2008.21.2514. Epub 2009 Oct 5. PMID 19805687
- [Background] Arico M, Schrappe M, Hunger SP, Carroll WL, Conter V, Galimberti S, Manabe A, Saha V, Baruchel A, Vettenranta K, Horibe K, Benoit Y, Pieters R, Escherich G, Silverman LB, Pui CH, Valsecchi MG. Clinical outcome of children with newly diagnosed Philadelphia chromosome-positive acute lymphoblastic leukemia treated between 1995 and 2005. J Clin Oncol. 2010 Nov 1;28(31):4755-61. doi: 10.1200/JCO.2010.30.1325. Epub 2010 Sep 27. PMID 20876426
- Available data/document: Individual Participant Data Set: CAMS-Ph+B-ALL — https://login.imedidata.com — CAMS-Ph+ALL-2025 DATASET